CLINICAL TRIAL: NCT07095790
Title: Tirofiban With Sequential Dual Antiplatelet Therapy Versus Dual Antiplatelet Therapy Alone in Mild Acute Ischemic Stroke (TiMIS): A Multicenter, Open-Label, Blinded-Endpoint, Parallel-Controlled, Randomized Clinical Trial
Brief Title: Tirofiban With Sequential Dual Antiplatelet Therapy in Mild Stroke
Acronym: TiMIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK2025063; 2024yb48 (Other Grant/Funding Number: Scientific research project of Xi'an Health Commission)
Record Dates: First submitted 2025-07-13; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mild Stroke
Keywords: Tirofiban; Dual Antiplatelet Therapy; Mild Stroke
MeSH Terms: interventions — Tirofiban; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban+Oral Dual Antiplatelet Therapy (Experimental): Patients will receive tirofiban in the first 48 hours and then be switched to oral dual antiplatelet therapy thereafter
  Interventions: Drug: Tirofiban+Oral Dual Antiplatelet Therapy
- oral dual antiplatelet therapy (Active Comparator): Patients will receive oral dual antiplatelet therapy alone
  Interventions: Drug: Oral Dual Antiplatelet Therapy

INTERVENTIONS:
Drug: Tirofiban+Oral Dual Antiplatelet Therapy — Tirofiban will use a loading dose, 0.4 μg/kg/min × 30 minutes, then 0.1μg/kg/min infusion for 47.5 hours; sequential Oral Dual Antiplatelet Therapy (Aspirin 100mg qd; Clopidogrel 75mg qd)
  Other Names: Tirofiban with Sequential Dual Antiplatelet Therapy
  Arms: Tirofiban+Oral Dual Antiplatelet Therapy
Drug: Oral Dual Antiplatelet Therapy — Aspirin 100mg qd; Clopidogrel 75mg qd (after first dose of 300mg)
  Other Names: Dual Antiplatelet Therapy; Aspirin plus Clopidogrel
  Arms: oral dual antiplatelet therapy

SUMMARY:
This study aims to evaluate whether initiating intravenous tirofiban within 48 hours of onset (with a 48-hour infusion), followed by sequential DAPT, can improve the likelihood of excellent functional outcomes (modified Rankin Scale score 0-1) in mild stroke patients, compared with standard DAPT therapy based on current guidelines.

DETAILED DESCRIPTION:
Although dual antiplatelet therapy (DAPT) reduces stroke recurrence and disability risks, its efficacy is limited in patients with mild ischemic stroke (NIHSS ≤5), among whom early neurological deterioration (END) and poor functional outcomes are frequently observed. Notably, intravenous thrombolysis is not more effective than DAPT for mild stroke management. Tirofiban, a glycoprotein IIb/IIIa receptor inhibitor, has shown potential efficacy in mild-to-moderate ischemic stroke, but robust evidence specific to mild stroke remains lacking. This study aims to evaluate whether initiating intravenous tirofiban within 48 hours of onset (with a 48-hour infusion), followed by sequential DAPT, can improve the likelihood of excellent functional outcomes (modified Rankin Scale score 0-1) in mild stroke patients, compared with standard DAPT therapy based on current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old.
2. Acute mild non-cardioembolic stroke.
3. NIHSS score ≤5.
4. Time from onset to randomization of ≤48 hours; if the time of onset is unknown, time from the last known time of being well to randomization of ≤48 hours.
5. The investigational drug can be administered within 48 hours of symptom onset.
6. Signed informed consent by the patient or legally authorized representative.

Exclusion Criteria:

1. Received or planned to receive intravenous thrombolysis or bridging therapy (with subsequent endovascular treatment)
2. Intracranial hemorrhage confirmed by imaging.
3. Pre-stroke modified Rankin Scale (mRS) score ≥2.
4. Any confirmed cardioembolic source, including chronic or paroxysmal atrial fibrillation, sick sinus syndrome, mitral stenosis, mechanical heart valve, infective endocarditis, intracardiac thrombus or vegetation, myocardial infarction within 3 months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction <30%.
5. History of primary intracerebral hemorrhage.
6. History of other intracranial hemorrhage (intraventricular, subarachnoid, epidural, or subdural hemorrhage).
7. Untreated or inadequately treated intracranial aneurysm or vascular malformation.
8. Major systemic bleeding within 30 days.
9. Active bleeding, including laboratory evidence of coagulopathy (platelet count <100 × 10⁹/L, activated partial thromboplastin time >50 seconds, or international normalized ratio >1.7), or treatment with direct oral anticoagulants within the preceding 48 hours.
10. Major surgery within 14 days.
11. Persistently elevated blood pressure (systolic >180 mmHg or diastolic >110 mmHg) despite treatment.
12. Baseline platelet count <100 × 10⁹/L.
13. Severe renal dysfunction (glomerular filtration rate <30 mL/min or serum creatinine >220 μmol/L [2.5 mg/dL]).
14. Known allergy or contraindication to tirofiban or aspirin.
15. Current pregnancy or lactation.
16. Any intracranial tumor (except asymptomatic meningiomas ≤1.5 cm in diameter).
17. Any terminal illness with life expectancy <6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of excellent functional outcomes (mRS 0-1) | 90 days
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death)

SECONDARY OUTCOMES:
Incidence of early neurological deterioration | 72 hours
  more than 2 National Institutes of Health Stroke Scale score increase (not result of cerebral hemorrhage) compared with baseline. National Institutes of Health Stroke Scale: stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms.
Incidence of early neurological improvement | 72 hours
  National Institutes of Health Stroke Scale score of 0 or improvement ≥2 points from baseline. National Institutes of Health Stroke Scale: stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms
Change in National Institutes of Health Stroke Scale score from baseline | 7 days
  National Institutes of Health Stroke Scale: stroke symptom severity scale with a range of 0-42. Higher score means more severe stroke symptoms
Proportion of good functional outcomes (mRS 0-2) | 90 days
  good functional outcomes (mRS 0-2)
Distribution of mRS scores | 90 days
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death)
Incidence of schemic stroke | 90 days
  new schemic stroke
Incidence of major adverse cardiovascular events | 90 days
  including ischemic stroke, hemorrhagic stroke, transient ischemic attack, myocardial infarction, and vascular death
Rate of symptomatic intracerebral hemorrhage | 7 days
  Symptomatic intracranial hemorrhage is defined according to the ECASS Classification
Rate of all-cause mortality | 90 days
  The mRS is an ordinal, graded interval scale that assigns patients among 7 global disability levels, which ranging from 0 (no symptom) to 5 (severe disability) and 6 (death).
Rate of major bleeding events | 90 days
  defined by the GUSTO bleeding criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Shi, M.D, Principal Investigator — Second Affiliated Hospital of Soochow University
Locations (18):
- China (18):
  - Suzhou Municipal Hospital of Anhui Province, Suzhou, Anhui
  - Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Taikang Xian People's Hospital, Zhoukou, Henan
  - WuYuan County People's Hospital, Bayan Nur, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Jiangsu Province (Suqian) Hospital, Suqian, Jiangsu
  - Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Jiangsu Shengze Hospital of Nanjing Medical University, Suzhou, Jiangsu
  - Changshu No.1 People's Hospital, Suzhou, Jiangsu
  - First People's Hospital of Kunshan, Suzhou, Jiangsu
  - Suzhou Ninth People's Hospital, Suzhou, Jiangsu
  - Suzhou Xiangcheng People's Hospital, Suzhou, Jiangsu
  - Taicang TCM Hospital Affiliated to Nanjing University of Chinese Medicine, Suzhou, Jiangsu
  - Zhangjiagang Hospital of Traditional Chinese Medicine, Suzhou, Jiangsu
  - Taixing Second People's Hospital, Taizhou, Jiangsu
  - Nuclear Industry 417 Hospital, Xi'an, Shaanxi
  - First People's Hospital of Xianyang, Xianyang, Shaanxi
  - Second Hospital of Tianjin Medical University, Tianjin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT07095790/SAP_000.pdf